CLINICAL TRIAL: NCT00555269
Title: Comparison of Macular Function and Visual Fields After Membrane Blue or Infracyanine Green Staining in Vitreoretinal Surgery
Brief Title: Membrane Blue Versus Infracyanine Green
Status: Completed | Type: Observational
Sponsor: The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery (Other)
Responsible Party: Univ.Prof.Dr. Susanne Binder, Ludwig Boltzmann Institute for Retinology and Biomicroscopic Lasersurgery
Other Study IDs: MB vs IFCG
Record Dates: First submitted 2007-11-07; First posted 2007-11-08 (Estimated); Last update posted 2009-04-22 (Estimated); Status verified 2009-04

CONDITIONS: Macular Pucker; Macular Hole
Keywords: Macular pucker; Macular hole; Membrane Blue; Infracyanine Green; Peripheral Visual Field
MeSH Terms: conditions — Epiretinal Membrane; Retinal Perforations

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MB
- IFCG

SUMMARY:
To compare possible toxicities of membrane blue and infracyanine green in vivo by macular function and peripheral visual field.

ELIGIBILITY:
Inclusion Criteria:

* Macular pucker or macular hole

Exclusion Criteria:

* Any other retinal disease

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a macular pucker or a macular hole, without any other retinal disease
Enrollment: 30 (Actual)
Dates: Start 2004-10; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Visual acuity, macular thickness and peripheral visual field

CONTACTS AND LOCATIONS:
Overall Officials: Katharina E Schmid-Kubista, MD, Principal Investigator — Ludwig Boltzmann Institute for Retinology and Biomicroscopic Lasersurgery

REFERENCES:
- [Derived] Schmid-Kubista KE, Lamar PD, Schenk A, Stolba U, Binder S. Comparison of macular function and visual fields after membrane blue or infracyanine green staining in vitreoretinal surgery. Graefes Arch Clin Exp Ophthalmol. 2010 Mar;248(3):381-8. doi: 10.1007/s00417-009-1213-4. Epub 2009 Oct 13. PMID 19823863